CLINICAL TRIAL: NCT02513342
Title: Endostar First-line Treatment of Advanced Non-small Cell Lung Squamous Carcinoma Based on Chemotherapy for Advanced Non-small Cell Lung Squamous Carcinoma Patients：a Randomized Controlled,Open, Multicenter Clinical Study
Brief Title: Endostar First-line Treatment of Advanced Non-small Cell Lung Squamous Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing NingQi Medicine Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSLCG-001
Record Dates: First submitted 2015-07-17; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-03

CONDITIONS: Advanced Lung Squamous Carcinoma
Keywords: Endostar,Advanced lung squamous carcinoma
MeSH Terms: interventions — endostar protein; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endostar+Docetaxel+Cisplatin (Experimental): Patients in this group will be given conventional chemotherapy medicine: Docetaxel+Cisplatin chemotherapy recommended by treatment guidelines for Advanced Non-small Cell Lung Squamous Carcinoma , and the Endostar-Recombinant human endostatin injection is injected by 30mg continuous intravenous injection pump,d1-d7.
  Interventions: Biological: Endostar; Drug: Docetaxel; Drug: Cisplatin
- Docetaxel+Cisplatin (Active Comparator): Patients in this group will be given conventional chemotherapy medicine: Docetaxel+Cisplatin chemotherapy recommended by treatment guidelines for Advanced Non-small Cell Lung Squamous Carcinoma.
  Interventions: Drug: Docetaxel; Drug: Cisplatin

INTERVENTIONS:
Biological: Endostar — Endostar 30mg continuous intravenous injection pump,d1-d7；
  Arms: Endostar+Docetaxel+Cisplatin
Drug: Docetaxel — d4 Docetaxel，75（mg/m2），iv；
Drug: Cisplatin — d4，cisplatin，75（mg/m2），iv；

SUMMARY:
Explore the efficacy and safety of the treatment of Endostar continuous intravenous injection pump combined DP scheme for first-line advanced lung squamous carcinoma and maintenance treatment., and explore the predicted biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Cytological and histological confirmation（Do not accept single sputum cytology in the diagnosis of patients） in patients diagnosed of lung squamous carcinoma;
2. According to a new IASLC2009 lung cancer TNM stages judged stage IIIB or IV non-small cell lung cancer.
3. Must have at least one evaluated lesion,according to the RRECIST version 1.1 standard (the longest diameter on spiral CT at least 10 mm,the longest diameter on plain CT at least 20 mm);
4. Male or female, age between 18 and 75 years old ;
5. ECOG PS 0~1；
6. Expected survival period ≥ 3 months or more
7. Enough blood function: absolute neutrophil count (ANC)≥2 x 109 / L and the platelet count≥ 100 x 109 / L and hemoglobin ≥9 g/dL;
8. Enough liver function: total bilirubin acuities≤the upper limit of normal (ULN); AST and ALT acuities ≤2.5 times of the upper limit of normal (ULN); Alkaline phosphatase ≤5 times of the upper limit of normal(ULN);
9. Enough renal function：serum creatinine ≤the limit of normal(ULN) or calculated creatinine clearance≥60 mL/min.
10. The electrocardiogram (ecg) basicaly normal,the body had no to heal wounds
11. No previous anti-tumor drug therapy, or only received for non metastatic tumor of adjuvant or neoadjuvant chemotherapy, but has ended more than six months before the study start.
12. Patients had surgery before,but have more than 4 weeks before the study star, and the patient has recovered;
13. Women with cmpleted uterus before intact in the group within 28 days must have a negative pregnancy test results (unles amenorrhea for 24 months). If the pregnancy test from the first time for more than 7 days,the patients need for urine pregnancy test(within 7 days before the first delivery).
14. Prior to biological agents, especially e. coli genetically engineered products without severe allergic reactions;
15. Sign the informed consent.

Exclusion Criteria:

1. Pregnancy, nursing mothers, or female patients with fertility but no contraception.
2. Existing serious acute infection, and can not be controlled; Or with fester sex and chronic infection,or wound in delay;
3. Original serious heart disease, including: congestive heart failure, uncontroled high risk arrhythmia, unstable angina, myocardial infarction, severe valvular heart disease, and resistant hypertension;
4. With uncontroled nerve, mental illness or mental disorders, compliance is poor, can't cooperate and response to treatment; Uncontroled primary brain tumors or CNS metastases illness, with obvious symptoms in cranial hypertension or nerve spirit;
5. With a bleeding tendency
6. Researchers believe that patients should not participate in this test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to month 36
  FS is a tumor progression or death time of a patient who has an objective record on the date of enrollment. PFS calculation end if the patient was lost, unknow death , or other anti tumor therapy was used.

SECONDARY OUTCOMES:
overall remission rate(ORR) | change from Baseline at the week 6, 12 of the treatment phase, the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase.
Disease control rate （DCR） | change from Baseline at the week 6, 12 of the treatment phase, the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase.
Overall survival（OS） | change from Baseline at the week 6, 12 of the treatment phase, the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jinling Hospital, Nanjing, Jiangsu
  - The first affiliated hospital of soochow university, Suzhou, Jiangsu